CLINICAL TRIAL: NCT06594237
Title: Maternal And Fetal Outcomes in Pregnant Women With Liver Disease
Status: Completed | Type: Observational
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Other Study IDs: NishterMultan-2
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fulminant Hepatic Failure
MeSH Terms: conditions — Liver Failure, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver disease complications during pregnancy can impact maternal and neonatal health, though not many studies are on view to investigate maternal and fetal outcomes in Pakistani pregnant women. So, this study was aimed to determine the maternal and fetal outcomes among pregnant females with liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females with liver disease
* With gestational age > 24 weeks
* Any parity or gravidity status

Exclusion Criteria:

* Pregnant females with renal disease or any kind of malignancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant females with gestational age > 24 weeks, regardless of their parity or gravidity status, with liver disease were enrolled in this study. Those with renal disease or any kinds of malignancy were not part of the study.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Maternal or Fetal survival or mortality. | 24 hours
  Fetal and maternal outcomes in terms of survival or death were noted.

CONTACTS AND LOCATIONS:
Overall Officials: Mehnaz Khakwani, FCPS, Principal Investigator — Department of Obstetrics & Gynecology, Nishtar Hospital, Multan; Hajra Sultana, FCPS, Principal Investigator — Department of Obstetrics & Gynecology, Nishtar Hospital, Multan
Locations (1):
- Nishtar Medical University, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared with other researchers on a reasonable request.